CLINICAL TRIAL: NCT00183677
Title: Biochemical Brain Changes Correlated With the Antidepressant Effect of Escitalopram: A Magnetic Resonance Spectroscopic Imaging Study
Brief Title: Brain Energy Metabolism in Individuals With Major Depressive Disorder Receiving Escitalopram
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David Mischoulon, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23MH067111 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Depression
Keywords: Brain Bioenergetic Metabolism; Magnetic Resonance Spectroscopy; Major Depressive Disorder; Treatment Response
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escitalopram (Experimental): Participants will receive open treatment with escitalopram.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10 to 30 mg per day for 12 weeks
  Other Names: Lexapro

SUMMARY:
This study will evaluate changes in brain energy metabolism due to treatment with escitalopram in people with major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a severe form of depression. MDD can significantly interfere with an individual's thoughts, behavior, mood, and physical health. People who suffer from MDD often experience feelings of worthlessness; they may feel hopeless and may be unable to cope with problems in their life. In addition, they often experience sleep disruption, loss of appetite, and chronic pain.

Antidepressant medications are often prescribed for treating MDD; however, 30% to 40% of individuals fail to respond adequately to medication. Preliminary research has shown that lower levels of brain energy metabolism are often associated with MDD. No studies have yet shown whether there is a difference in brain energy metabolism between individuals who respond well to antidepressants versus those who do not. Escitalopram is an antidepressant medication often used to treat MDD. It causes a calming effect and reduces anxiety by increasing the amount of serotonin in the brain. This study will compare the changes in brain energy metabolism due to treatment with escitalopram in individuals with MDD. In turn, these findings may aid in understanding the relationship between brain energy metabolism and depression, and may guide future antidepressant trials.

This 12-week study will enroll individuals diagnosed with MDD, as well as healthy individuals. During Weeks 1 through 4, participants with MDD will receive 10 mg of escitalopram on a daily basis. If a participant does not respond well to the medication, as determined by the study clinician, the dose may be increased to 20 mg per day for Weeks 5 through 8. If a participant continues to not respond to the medication after 8 weeks, the dose may be increased to 30 mg per day for Weeks 9 through 12. Study visits will occur every other week throughout the 12 weeks. Laboratory tests, physical examinations, and vital sign measurements will be performed at each study visit. Outcome measurements will include depression levels as assessed by standardized psychological tests and questionnaires, as well as brain energy metabolite levels as assessed by magnetic resonance spectroscopy (MRS) and magnetic resonance imaging (MRI) scans. The MRS and MRI scans will occur at baseline, Week 2, and Week 12; the entire scanning procedure will last 70-80 minutes. Following the end of the study, all participants will be offered follow-up medical care for 3 months. Participants who responded well to escitalopram will be offered continued treatment with the drug, while those who did not respond well to escitalopram will be offered treatment with another antidepressant.

ELIGIBILITY:
Inclusion Criteria:

For depressed subjects:

* Meets DSM-IV diagnostic criteria for major depressive disorder
* Score of greater than 16 on the Hamilton Depression Rating scale (17 items) at study entry
* Agrees to use an effective form of contraception throughout the study

For healthy volunteers:

* Not currently taking any medications
* No lifetime history of major neurological, medical, psychiatric disorder, or head injury
* Agrees to use an effective form of contraception throughout the study

Exclusion Criteria:

* Current suicidal ideation that may make study participation unsafe
* Current serious or unstable medical illness (e.g., cardiovascular, kidney, liver, respiratory, endocrine, neurologic, or blood-related disease)
* History of seizure disorder
* History of or current DSM-IV diagnosis of any of the following psychiatric illnesses within 12 months of study entry: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, mood congruent or mood incongruent psychotic features, substance dependence disorders (including alcohol)
* History of or current diagnosis of dementia, or a score of less than 26 on the Mini Mental Status Examination at screening
* History of multiple adverse drug reactions or allergic reaction to the study drugs
* Currently taking psychotropic drugs or antidepressant medications
* Clinical or laboratory evidence of hypothyroidism
* Failure to respond during current major depressive episode to at least one adequate antidepressant trial, defined as 6 weeks or more of treatment with 40 mg of citalopram per day (or its antidepressant equivalent)
* History of electroconvulsive therapy (ECT) within the 6 months prior to study entry
* Pregnant
* Subjects with a CGI score a 6 ("severely depressed") or 7 ("among the most extremely depressed patients")
* A BMI of 39 or greater, for comfort in scanner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2003-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan V. Iosifescu, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Escitalopram: Participants will receive treatment with escitalopram.
Period: Overall Study
Arm/Group | Open Label Escitalopram
Started | 97
Completed | 53
Not Completed | 44

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Escitalopram
Number analyzed (Participants) | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 97
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.54 (13.42)
Gender [Count of Participants; unit: Participants]
  Female | 42
  Male | 55
Region of Enrollment [Number; unit: participants]
  United States | 97

OUTCOME MEASURES:

1. Primary Outcome: Responder and Remission Status (%), Based on the Depression Rating Scale Score
Description: The Hamilton Depression Rating Scale, 17 items (HAMD-17, range 0-52) was used to measure changes in depression severity from baseline to endpoint. Clinical Responder status was defined as > 50% improvement (i.e., reduction) in HAMD-17 score from baseline to endpoint. Clinical Remission status was defined as HAMD-17 score < 8 at endpoint (week 12 visit).
Time Frame: Measured at Week 12
Population: 97 patients with MDD (42 Female) enrolled in the 12 week study, 53 patients (27 Female) completed. Only completers were included in the primary outcome measure.
Measure: Number; unit: participants
Groups:
- Open Label Escitalopram: Participants received open treatment with escitalopram.
Arm/Group | Open Label Escitalopram
Number analyzed (Participants) | 53
participants
  Clinical Responders | 36
  Clinical Remitters | 32

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 12 weeks of participation in the study.
Description: All gastrointestinal symptoms (e.g., nausea, diarrhea) were collected under the category gastrointestinal upset ("GI upset")
Arm/Group | Open Label Escitalopram
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 45/97
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Escitalopram (N=97)
Fatigue (Psychiatric disorders) | 23 (23) — Fatigue includes report of fatigue, sedation, drowsiness, hypersomnia, and/or lethargy.
GI Upset (Gastrointestinal disorders) | 17 (17) — GI upset includes report of GI upset, nausea, diarrhea, gas, stomach cramps, and/or indigestion
Headache (General disorders) | 11 (11)
Insomnia/Sleep Disturbance (General disorders) | 11 (11)
Sexual Side Effects (Reproductive system and breast disorders) | 10 (10) — Sexual side effects include report of decreased sexual drive, anorgasmia, or erectile dysfunction.
Agitation (Psychiatric disorders) | 6 (6) — Agitation includes report of agitation, jitteriness, and internal restlessness.
Decreased Appetite (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No